CLINICAL TRIAL: NCT02402764
Title: Investigator-Initiated Phase 2 Clinical Trial of Selinexor (KPT-330) for the Treatment of Metastatic Triple Negative Breast Cancer
Brief Title: Phase 2 Trial of Selinexor (KPT-330) for Metastatic Triple Negative Breast Cancer (TNBC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18150
Record Dates: First submitted 2015-03-25; First posted 2015-03-30 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer
Keywords: Triple Negative Breast Cancer (TNBC); Breast - Female; Breast - Male; Metastatic Triple Negative Breast Cancer; Receptor Tyrosine-protein Kinase erbB-2 (HER2) Negative; Erythroblastosis virus oncogene B (erbB)
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Selinexor Treatment (Experimental): Screening period (which may last up to 28 days), followed by Selinexor treatment for qualified participants.
  During the treatment period, participants will undergo physical examination every 2 weeks until Cycle 6 Day 1 (C6D1), and then every 4 weeks and assessment of tumor response every 8 weeks.
  Participants will be treated until progression of disease or the development of unacceptable toxicities. All participants will then undergo a final visit (end of treatment visit).
  Interventions: Drug: Selinexor

INTERVENTIONS:
Drug: Selinexor — Participants will receive selinexor twice weekly on Monday/Wednesday, Tuesday/Thursday or Wednesday/Friday of Weeks 1, 2 and 3 of each 4-week cycle. Selinexor will not be taken during Week 4. One cycle is defined as 28 days or 6 doses. The starting dose for this trial is 60 mg (flat dose as long as their dose-based body surface area (BSA) analysis does not exceed 70 mg/m^2).
  Other Names: KPT-330; Selective Inhibitor of Nuclear Export (SINE)

SUMMARY:
The main purpose of this study is to see whether the combination of selinexor (KPT-330) can help people with triple negative breast cancer (TNBC). Researchers also want to study the safety and tolerability of Selinexor in TNBC patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed triple negative breast cancer (TNBC), defined as negative immunohistochemical staining for estrogen and progesterone receptors (≤5% of nuclei positive by IHC) and receptor tyrosine-protein kinase erbB-2 (HER2) negative (IHC 0-1+ or HER2-neu negative according to American Society of Clinical Oncology; College of American Pathologists (ASCO-CAP) HER2 Test Guideline Recommendations)
* Written informed consent in accordance with federal, local, and institutional guidelines
* Body surface area ≥1.4 m^2
* Age ≥18 years
* Estimated life expectancy of >3 months at study entry
* TNBC must be either locally recurrent or metastatic. Locally recurrent disease must not be amenable to surgical resection or radiation with curative intent.
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Documented disease progression at study entry
* Must have received at least 1 chemotherapy regimens in the setting of metastatic disease
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤2
* Adequate hematological function: Absolute neutrophil count (ANC) > 1500/mm^3, platelets count >100,000mm^3
* Adequate hepatic function within 14 days prior to Cycle 1 Day 1 (C1D1): total bilirubin <2 times the upper limit of normal (ULN) (except patients with Gilbert's syndrome who must have a total bilirubin of < 3 times ULN) and aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤2.5 x ULN. In the case of known (radiological and/or biopsy documented) liver metastasis, AST/ALT ≤5.0 times ULN is acceptable.
* Amylase and lipase ≤ 1.5 x ULN
* Adequate renal function within 14 days prior to C1D1: estimated creatinine clearance of ≥ 30 mL/min
* Women of child-bearing potential (WOCBP) must agree to use dual methods of contraception and have a negative serum pregnancy test at screening, and male participants must use an effective barrier method of contraception if sexually active with a female of child-bearing potential. For both male and female participants, effective methods of contraception must be used throughout the study and for 3 months following the last dose. To be considered of non-childbearing potential, postmenopausal women must be amenorrheic for at least 12 months naturally (not in the setting of post chemotherapy) or participants must be surgically sterile.
* Must have received prior anthracycline and taxane therapy unless clinically contraindicated

Exclusion Criteria:

* Significant medical illness that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the participant's ability to tolerate this therapy
* Women who are pregnant or lactating
* Radiation, chemotherapy, or immunotherapy or any other approved anticancer therapy ≤2 weeks prior to cycle 1 day 1
* Major surgery within 4 weeks before Day 1
* Unstable cardiovascular function: Electrocardiogram (ECG) abnormalities requiring treatment, or congestive heart failure (CHF) of New York Hearth Association (NYHA) Class ≥3; myocardial infarction (MI) within 3 months
* Uncontrolled infection requiring parenteral antibiotics, antivirals, or antifungals within one week prior to first dose. Potential participants with controlled infection or on prophylactic antibiotics are permitted in the study.
* Known history of HIV
* Known active hepatitis A, B, or C infection that requires treatment
* Any underlying condition that would significantly interfere with the absorption of an oral medication
* Grade >2 peripheral neuropathy at baseline (within 14 days prior to cycle 1 day 1)
* Participation in an investigational anti-cancer study within 3 weeks prior to Cycle 1 Day 1
* Coagulation problems and active major bleeding within 4 weeks prior to C1D1 (peptic ulcer, epistaxis, spontaneous bleeding)
* Active central nervous system (CNS) malignancy. Asymptomatic small lesions are not considered active. Treated lesions may be considered inactive if they are stable for at least 3 months.
* Radiation, chemotherapy, or immunotherapy or any other anticancer therapy ≤ 2 weeks prior to Cycle 1 Day 1 or radio-immunotherapy ≤ 4 weeks prior to Cycle 1 Day 1
* Have not recovered to Grade ≤ 1 or to their baseline from clinically significant adverse effects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-07-08 (Actual); Primary Completion 2016-03-10 (Actual); Study Completion 2019-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyo S. Han, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Shafique M, Ismail-Khan R, Extermann M, Sullivan D, Goodridge D, Boulware D, Hogue D, Soliman H, Khong H, Han HS. A Phase II Trial of Selinexor (KPT-330) for Metastatic Triple-Negative Breast Cancer. Oncologist. 2019 Jul;24(7):887-e416. doi: 10.1634/theoncologist.2019-0231. Epub 2019 Apr 17. PMID 30996012

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at Moffitt Cancer Center between July 2015 and January 2016.
Groups:
- Selinexor Treatment: Ten patients were treated with oral selinexor 60 mg twice per week (on days 1 and 3) on a schedule of 3 weeks on and 1 week off, each four-week cycle.
Period: Overall Study
Arm/Group | Selinexor Treatment
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants
Arm/Group | Selinexor Treatment
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: years] | 60 [44 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate
Description: Complete Response (CR) + Partial Response (PR) + Stable Disease (SD) ≥ 12 weeks of selinexor in patients with triple negative breast cancer (TNBC), according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. CR: Disappearance of all target lesions; PR: At least a 30% decrease in the sum of the diameter (LD) of target lesions, taking as reference the baseline sum LD; Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Up to 10 months
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | Selinexor Treatment
Number analyzed (Participants) | 10
Participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 3
  Progressive Disease | 7

2. Secondary Outcome: Best Overall Response (OR)
Description: The best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The patient's best response assignment will depend on the achievement of both measurement and confirmation criteria.
Time Frame: Up to 10 months
Population: Participants with Complete Response or Partial Response
Arm/Group | Selinexor Treatment
Number analyzed (Participants) | 0

3. Secondary Outcome: Duration of Overall Response
Description: The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started) or death. The duration of overall CR is measured from the time measurement criteria are first met for CR until the first date that recurrent disease is objectively documented or death.
Time Frame: Up to 10 months
Population: Participants with Complete Response or Partial Response
Arm/Group | Selinexor Treatment
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: Median time to progression. Progression-free survival is defined as time elapsed from the beginning of study treatment to the first documentation of radiologic progression as defined by standard RECIST criteria or death.
Time Frame: Up to 10 months
Population: All participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Selinexor Treatment
Number analyzed (Participants) | 10
months | 1.0 [0.5 to 4.0]

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival, defined as the time from randomization to death from any cause.
Time Frame: End of post-treatment 12 month follow-up, up to 24 months per participant
Population: All participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Selinexor Treatment
Number analyzed (Participants) | 10
months | 6.0 [1.7 to 10.4]

ADVERSE EVENTS:
Time Frame: 10 months
Arm/Group | Selinexor Treatment
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selinexor Treatment (N=10)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selinexor Treatment (N=10)
Constipation (Gastrointestinal disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 4 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Platelet count decreased (Investigations) | 3 (6)
Alanine aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (2)
Investigations - Other, specify (Investigations) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blurred vision (Eye disorders) | 4 (4)
Fatigue (General disorders) | 3 (5)
Fever (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Irritability (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Hot flashes (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes